CLINICAL TRIAL: NCT03500575
Title: Extracorporeal Photopheresis as Induction Therapy to Prevent Acute Rejection After Lung Transplantation in Cystic Fibrosis Patients
Brief Title: Extracorporeal Photopheresis in Lung Transplant Rejection for Cystic Fibrosis (CF) Patients
Acronym: PHORLUCY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Italian Cystic Fibrosis Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1708
Record Dates: First submitted 2018-03-02; First posted 2018-04-18 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Lung Transplant Rejection
Keywords: induction therapy, photopheresis
MeSH Terms: interventions — Photopheresis

STUDY DESIGN:
Intervention Model Description: Pilot study, single center, randomized controlled trial, single blind, 2 parallel arms
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- photopheresis (Experimental)
  Interventions: Device: photopheresis
- control (No Intervention)

INTERVENTIONS:
Device: photopheresis — • Treated group will receive ECP with Therakos online system. Each session consists in 1 treatment for 2 consecutive days. First session stars within 72 hours after transplantation followed by a session weekly for 3 time and 2 sessions for the next 2 months (6 sessions = 12 treatment)
  Arms: photopheresis

SUMMARY:
Background/Rationale Acute rejection (AR) is common in the first year after lung transplantation. AR has usually been reversible with treatment, but it can trigger chronic rejection that is the leading causes of late morbidity and mortality. Extracorporeal photopheresis (ECP) has emerged as a promising treatment for chronic rejection. The investigators postulate that the immunoregulatory property of ECP could promote graft tolerance immediately after lung transplantation.

Objectives The aim of this trial is to evaluate the safety and efficacy of ECP as induction therapy for prevention of AR in recipients affected with cystic fibrosis in the first year after lung transplantation. The extracellular vesicles in the cell-to-cell communication and immunomodulation will be also investigated.

Preliminary results (personal) A preliminary study, conducted in Vienna, demonstrated that 9 patients treated with ECP as induction therapy had 0% of chronic rejection versus 50% in the control group. The Institution hosting the current project is among largest lung transplantation centers in Italy with high rate of cystic fibrosis recipients. The Institution has experience in ECP and a dedicated instrument was specifically bought for the project. Internal collaborators have strong expertise in biological aspects including the extracellular vesicle compartment.

DETAILED DESCRIPTION:
The aim of this pilot trial is evaluate the efficacy and safety of ECP as induction therapy for prevention of AR in recipients affected of cystic fibrosis in the first year after lung transplantation.

The investigators postulate that ECP could induce graft immunotolerance avoiding the development of chronic rejection. Exposing T-cells to ultraviolet light results in DNA damage and apoptosis; such form of cell death does not typically stimulate a prolonged inflammatory cascade. When re-infused to the patient, apoptotic T-cells are surrounded by antigen presenting cells (APCs). The large number of APCs encircling the damaged T-cells limits the inflammatory response and stimulates specific signalling cascades in APCs that result in anti-inflammatory cytokine production; finally, immature dendritic cells could gain tolerogenic phenotypes. Based on this process, a theory postulates that the immuno-modulation secondary to ECP is related to a general increase in regulatory T-cells that cause a down-regulation of immune responses involved in chronic rejection onset. Another theory assumes that suppressor T-cells may acquire anti-clonal immunity prompted by the APCs; therefore, a sort of T-cell vaccination is the result of leukocyte apoptosis. The intention is to use this T-cell regulation to induce immunotolerance toward the graft before the development of chronic rejection, in spite to operate when the damage is in progress. To activate this effect from the first hours after transplantation, it can be useful the immunomodulatory activity of extracorporeal photopheresis, already established by clinical studies applied to the treatment of acute and chronic rejection.

The efficacy of ECP as induction therapy will be measured with the identification of AR rate in the study group versus the control group. AR is diagnosed with trans-bronchial biopsy and graded using standard histological criteria: A0 (none), A1 (minimal), A2 (mild), A3 (moderate) or A4 (severe). A stable 10% decrease of forced expiratory volume in 1 second (FEV1) on baseline will be considered as AR even though trans-bronchial biopsy is not available. In addition, lymphocyte immunophenotype (with particular regard to CD4 + and CD25 +), the cytokine profile (interleukine (IL) 4, IL-10, IL-12 measured by High Resolution Cytokines Array) and the extracellular vesicles content are tested to assess the therapeutic response. Finally, anti-HLA antibodies are tested to understand their dynamics.

The ECP safety is assessed by recording every adverse effect with specific attention to opportunistic infections.

In conclusion, this study aims to verify whether the induction therapy with ECP can dramatically decrease the rate of acute rejection in order to impact positively on the main cause of mortality in lung transplantation: the chronic rejection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CF undergoing first lung transplantation
* Male or female
* Any ethnicity
* Patients must have a body weight more than 40 kg
* Patients must have a platelet count more than 20.000/cmm
* Patients must be willing of understanding the purpose and risks of the study and must sign a statement of informed consent
* Patients transplanted in the first year from the study beginning.

Exclusion Criteria:

* Previous organ transplantation
* Women who are pregnant and/or lactating
* Patients with hypersensitivity or allergy to both heparin and citrate products
* Patients who are unable to tolerate extracorporeal volume shifts associated with ECP treatment due to the presence of any of the following conditions:uncompensated congestive heart failure, pulmonary edema, renal failure or hepatic failure
* Patients who are transplanted following the Italian criteria for emergency transplantation.
* Patients who stay more than 72 hours in ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-05-20 (Estimated); Primary Completion 2021-12-10 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Acute Rejection (measure: number of events) | 36 months
  The diagnosis of acute rejection is done by transbronchial biopsy which are classified according the International Society of Heart and Lung Transplantation (ISHLT) grading. In alternative, the diagnosis of acute rejection is done by presence of one of the following clinical or radiological findings: reproducible decrease in lung function (FEV1), hypoxemia (pO2 < 60mmHg, Sao2< 90%), pulmonary infiltrates, pleural effusions or dyspnea without evidence of infection

SECONDARY OUTCOMES:
Infections from cytomegalovirus (CMV), bacteria, fungi, non-CMV virus, tuberculosis, parasitic (measure: number of events) | 12 months
  Bronchoscopy with microbiologic, bacteriology, mycology, virology, parasitology and tuberculosis investigation will be performed
overall survival | 12 months
  The overall survival will be registered in the first year after lung transplant. It will be reported as months to death and the cause of death
cumulative immunosuppressive therapy (measure: mg) | 12 months after transplant
  cumulative doses of Tacrolimus, azathioprine (AZT) and corticosteroids at 12 months
total hospitalization days after discharge (measure: days) | at 6 months and 12 months after primary discharge
  The average number of days spent in the hospital during the first year after transplant
freedom from chronic lung allograft disease (measure: months) | 12 months
  The efficacy of ECP as induction therapy will be measured with the identification of AR rate in the study group versus the control group. AR is diagnosed with trans-bronchial biopsy and graded using standard histological criteria: A0 (none), A1 (minimal), A2 (mild), A3 (moderate) or A4 (severe). A stable 10% decrease of forced expiratory volume in 1 second (FEV1) on baseline will be considered as AR even though trans-bronchial biopsy is not available
side effects of ECP (measure: number of events) | 3 months after the latest treatment with ECP
  The ECP safety is assessed by recording every adverse effect with specific attention to opportunistic infections
lymphocyte immunophenotype (measure: pg/ml) by cluster of differentiation (CD) | At time zero and 48 hours after the end of each sessions of two ECP treatments peripheral blood samples will be collected
  lymphocyte immunophenotype (CD45, CD3, CD19, CD14, CD56/16, CD4, CD8, HLA-DR (human leukocyte antigen D Related), CD16, CD25, CD127, CD11c, Annexin/PI)
cytokine profile of interleukyn (IL) (number/mmc; percentage) | At time zero and 48 hours after the end of each sessions of two ECP treatments peripheral blood samples will be collected
  the cytokine profile (IL-4, IL-10, IL-12 measured by High Resolution Cytokines Array) are tested to assess the therapeutic response.
extracellular vesicles content (measure: number/ml) | At time zero and 48 hours after the end of each sessions of two ECP treatments peripheral blood samples will be collected
  extracellular vesicles are important mediators of intercellular communication, being involved in the transmission of biological signals between cells. Number, membrane antigens, mRNA (messenger of ribonucleic acid) and protein content are tested. We use nanoparticle tracking analysis for the testing
anti-HLA antibodies profile (measure: µmg/ml) | At time zero, after 7 days of the end of each cycle of treatment, at 3, 6 months and one year after transplantation
  the anti-HLA antibodies will be tested by Luminex methodology

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz J, Winters JL, Padmanabhan A, Balogun RA, Delaney M, Linenberger ML, Szczepiorkowski ZM, Williams ME, Wu Y, Shaz BH. Guidelines on the use of therapeutic apheresis in clinical practice-evidence-based approach from the Writing Committee of the American Society for Apheresis: the sixth special issue. J Clin Apher. 2013 Jul;28(3):145-284. doi: 10.1002/jca.21276. PMID 23868759
- [Result] Aubin F, Mousson C. Ultraviolet light-induced regulatory (suppressor) T cells: an approach for promoting induction of operational allograft tolerance? Transplantation. 2004 Jan 15;77(1 Suppl):S29-31. doi: 10.1097/01.TP.0000112969.24120.64. PMID 14726767
- [Result] Durazzo TS, Tigelaar RE, Filler R, Hayday A, Girardi M, Edelson RL. Induction of monocyte-to-dendritic cell maturation by extracorporeal photochemotherapy: initiation via direct platelet signaling. Transfus Apher Sci. 2014 Jun;50(3):370-8. doi: 10.1016/j.transci.2013.11.008. Epub 2013 Nov 28. PMID 24360371
- [Derived] Righi I, Fenizia C, Trabattoni D, Nosotti M, Grisorio G, Vanetti C, di Tella S, Mocellin C, Fantini N, Prati D, Morlacchi LC, Rossetti V, Blasi F, Clerici M, Rosso LP. Extracorporeal photopheresis as induction therapy in lung transplantation for cystic fibrosis: a pilot randomized trial. Front Immunol. 2025 May 16;16:1583460. doi: 10.3389/fimmu.2025.1583460. eCollection 2025. PMID 40453071